CLINICAL TRIAL: NCT03814278
Title: A Pilot Randomized Controlled Trial On Complete Bed Rest Versus Activity Restriction After Preterm Premature Rupture of the Membranes
Brief Title: Bed Rest After Preterm Premature Rupture of the Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Lisboa Norte (Other)
Responsible Party: Principal Investigator, Inês Martins, Medical Doctor, Principal Investigator, Centro Hospitalar Lisboa Norte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RPM-PT_Estudo_Repouso
Record Dates: First submitted 2018-11-23; First posted 2019-01-24 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete bed rest (Experimental): Participants on complete bed rest group kept antepartum confinement to bed with toileting restricted to bedpan use. Participants in this group received prophylactic subcutaneous enoxaparin (40mg/day).
  Interventions: Behavioral: complete bed rest
- Activity restriction group (Experimental): Activity restriction group had motion limited to bathroom privileges and walks to the ward canteen four times per day.
  Interventions: Behavioral: activity restriction

INTERVENTIONS:
Behavioral: complete bed rest — Patients in this group received standard care for PPROM according to the institution protocol, including antepartum confinement to bed.
  Arms: Complete bed rest
Behavioral: activity restriction — Patients in this group received standard care for PPROM according to the institution protocol but to had bathroom privileges and walks to the ward canteen four times per day.
  Arms: Activity restriction group

SUMMARY:
Antepartum bed rest is widely prescribed after preterm premature rupture of the membranes (PPROM), although its effectiveness to prevent preterm birth has not been demonstrated. This pilot randomized controled trial (RCT) aims to access the impact of bed rest in maternal and neonatal outcomes in pregnancies complicated by premature rupture of the membranes.

DETAILED DESCRIPTION:
Aims - To access the impact of bed rest in latency time to delivery, chorioamnionitis incidence and other maternal and neonatal outcomes in pregnancies complicated by PPROM, thus enabling proper sample size calculation for future powered RCT.

Study population and Sample size - Eligible patients included those with single pregnancies with PPROM at 24+0-33+6 weeks of gestation who were admitted to and delivering at our tertiary center. PPROM was diagnosed on the basis of patient's history and sterile speculum examination with visualization of amniotic fluid pooling in the vagina and/or leaking from the cervical canal. Exclusion criteria included indication for immediate delivery on admission (chorioamnionitis, placenta abruption, cord prolapse, signs of fetal hypoxia/distress), fetal malformations, multiple gestation, and maternal immunosuppressive disease. Considering future sample size calculation based upon assumed differences between groups regarding latency and infection, we aimed a sample of 30 participants.

Randomization - A pilot unblinded randomized controlled trial (RCT) in a 1:1 allocation ratio between two groups (complete bed rest versus activity restriction after PPROM). Simple random allocation sequence was generated by the investigators and implemented by sequentially numbered sealed envelopes. Participants were enrolled by physicians after hospital admission and written informed consent was obtained before randomization. The trial was conducted in a single tertiary center of the Portuguese national health system after approval by its ethical committee.

Statistical analysis - An intention-to-treat analysis was performed with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancies AND
* PPROM at 24+0-33+6 weeks of gestation AND
* admitted to our tertiary center.

Exclusion Criteria:

* indication for immediate delivery on admission (chorioamnionitis, placenta abruption, cord prolapse, signs of fetal hypoxia/distress)
* fetal malformations
* multiple gestation
* maternal immunosuppressive disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patient eligibility is based on gender identity because we will include only pregnant women
Enrollment: 32 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Latency time | From preterm premature rupture of the membranes until delivery, estimated average time of one week
  Time between preterm premature rupture of the membranes and delivery, in days
Chorioamnionitis | From preterm premature rupture of the membranes until delivery, estimated average time of one week
  Incidence of clinical chorioamnionitis (defined as maternal fever plus leukocytosis and CRP elevation, or as maternal fever plus any two of the following: fetal tachycardia; maternal tachycardia; uterine tenderness; purulent amniotic fluid)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT03814278/Prot_SAP_000.pdf